CLINICAL TRIAL: NCT06290440
Title: Development of Medication Counselling Models for Outpatient Oral Anticoagulant-taking Patients
Brief Title: MEdication Counselling Models for Outpatient oRal antIcoaguLation
Acronym: MEMORIAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gia Dinh People Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 28/NDGD-HDDD
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Anticoagulants; Circulating, Hemorrhagic Disorder
Keywords: oral anticoagulant; counselling; distance counselling; medication adherence; knowledge; hospitalisation; mortality; venous thromboembolism
MeSH Terms: conditions — Hemorrhagic Disorders; Medication Adherence; Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist-led counselling (Active Comparator)
  Interventions: Other: Pharmacist-led counselling
- Telepharmacy-led counselling (Experimental)
  Interventions: Other: Telepharmacy-led counselling

INTERVENTIONS:
Other: Telepharmacy-led counselling — The counselling process will be delivered as follows: (1) researchers assist patients in signing up and using the telepharmacy application; (2) researchers send the counselling information from the telepharmacy application to the patient's account (the information will be provided as leaflets and 3-5-minute videos to improve the accessibility); (3) the integrated chatbot system forwards any additional questions or concerns of the patients to the counselling pharmacists; and (4) the pharmacists directly address the patient's questions or concerns through phone calls within the shortest possible timeframe.
  Arms: Telepharmacy-led counselling
Other: Pharmacist-led counselling — Pharmacists will counsel the patients on how to use their OAC. Each counselling section will take approximately 7-15 minutes, depending on the patient's questions or concerns. The counselling contents have already been compiled and validated by NDGD Hospital to ensure rationale and simplicity for every patient. Counselling pharmacists have received specialised training in drug information and patient communication so intervention delivery will be consistent across different pharmacists.
  Arms: Pharmacist-led counselling

SUMMARY:
The goal of this clinical trial is to investigate whether telepharmacy-led counselling can improve medication adherence, knowledge, and hospitalisation/mortality compared with pharmacist-led counselling in adult outpatients taking oral anticoagulants.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* taking oral anticoagulants
* using smartphones that can access the telepharmacy application
* agreeing to participate

Exclusion Criteria:

* pregnancy or lactation
* having cancer
* having immunodeficiency disorders or using immunosuppressants
* renal impairment (creatinine clearance <30 mL/min)
* hepatic impairment (Child-Pugh B or C cirrhosis)
* heart failure (class IV, New York Heart Association)
* history of myocardial infarction or stroke within the latest 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | Measured at month 1, 6, and 12 after randomisation
  Measured using Morisky-Green-Levine scale. The levels of adherence are: (1) high (0 point); (2) medium (1-2 points); and (3) low (3-4 points).

SECONDARY OUTCOMES:
Knowledge of oral anticoagulants | Measured at month 1, 6, and 12 after randomisation
  Measured using Anticoagulant Knowledge Tool scale that was modified and validated on Vietnamese patients. This includes two sections: (1) general knowledge of oral anticoagulants (16 questions with a maximum score of 21) and (2) specific knowledge of vitamin K antagonists (5 questions with a maximum score of 8, only for patients using vitamin K antagonists). For multiple-choice questions, 1 correct answer earns 1 point, while for short-answer questions, 1 correct answer may result in 1-3 points, depending on the questions. The standardized score will be presented as percentage (based on the maximum score of 21 for direct-acting oral anticoagulant-taking patients or 29 for those using vitamin K antagonists), with the higher score indicating better knowledge.
All-cause hospitalisation | 24 months after randomisation
  Measured using medical records and self-reported/family-reported information
VTE-related hospitalisation | 24 months after randomisation
  Measured using medical records and self-reported/family-reported information
Bleeding-related hospitalisation | 24 months after randomisation
  Measured using medical records and self-reported/family-reported information
All-cause mortality | 24 months after randomisation
  Measured using medical records and self-reported/family-reported information
VTE-related mortality | 24 months after randomisation
  Measured using medical records and self-reported/family-reported information
Bleeding-related mortality | 24 months after randomisation
  Measured using medical records and self-reported/family-reported information